CLINICAL TRIAL: NCT03578549
Title: Pulse Oximeter is a Potential Diagnostic Device for the Assessment of Pulpal Blood Flow
Brief Title: Diagnostic Device for the Assessment of Pulpal Blood Flow
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Darya Dabiri, Post Doc Research Fellow, Faculty of Anesthesiology, University of Michigan
Other Study IDs: HUM00136199
Record Dates: First submitted 2018-06-22; First posted 2018-07-06 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Dental Pulp Test
Keywords: Dental Pulp Test; Vitality Testing; Pulpal Blood Flow Measure
MeSH Terms: interventions — Oximetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Oximetry testing of healthy teeth and those requiring removal: To assess the ability of pulse oximeter to assess the presence of pulse in teeth and to correlate pulse oximeter readings with conventional pulp testing measures including cold test, electrical pulp test, percussion and palpation testings, pulse oximeter will be used with a special holding frame, for 15-30 seconds.
  Note: the reading will not affect clinical practice; it is simply to gather data to see if pulse oximetry can facilitate diagnostic practices in the future
  Interventions: Device: Pulse Oximetry

INTERVENTIONS:
Device: Pulse Oximetry — Pulse Oximeter is being applied with a special holding tool to test the oximeter for its ability to measure pulpal blood flow, but no effect of the oximeter is being measured. Thus, to that degree the use is observational rather than interventional.

SUMMARY:
The purpose of this study is to assess tooth health by using a pulse oximeter which measures the blood flow within the tooth. This method is not currently being used in dentistry. We hypothesize that if we can measure both sensation and blood flow in a tooth, we will be able to better determine if the tooth is "alive or dead". In the future, this method may help determine which teeth are diseased and require dental treatments.

DETAILED DESCRIPTION:
The vitality of the pulp is determined according to the health of the vascular supply not the sensory fibers. Conventional subjective tooth assessments (percussion, palpation, cold, and electrical pulp testing) and objective pulpal blood flow measurements will be used for teeth that are planned for extraction and also up to 2-5 additional teeth in each participant. The correlation between a single combined score from collective conventional subjective tooth assessments and the objective pulse oximetry reading for selected teeth will be used to evaluate if pulse oximeter measurements are a reliable marker for patient's reported symptoms.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, you must meet the following criteria:

1. Must be a patient of the Oral Surgery Clinic at the University of Michigan School of Dentistry
2. Must be scheduled for at least one tooth extraction at Oral Surgery Clinic
3. Must be able to understand and willing to cooperate with all study procedures
4. Must be able to sign an IRB-approved written consent
5. Must have at least two teeth with an intact crown, without any full metallic crown coverage, and/or previous root canal treatments
6. Must have no history of spontaneous pain, and/or lingering pain to cold/hot in teeth that are not going to be extracted on that day.
7. If one of the teeth mentioned in inclusion #6 is being extracted, be willing to give your extracted tooth/teeth for further analysis to determine of the tooth is "alive or dead"

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * If participant self-reports liver, kidney, heart, blood, metabolic or systemic disease which may make execution of the protocol or interpretation of the results difficult
  * If participant has severe physical impairments (e.g., complete blindness or deafness) and/or cognitive impairments (e.g., dementia) that precludes participation in the procedures outlined in this proposal
  * If participant is or could be pregnant
  * If participant is currently receiving radiation
  * If participant not able to hold mouth open for extended period of time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy individuals with 2-5 non-endodonticaly treated teeth in addition to the tooth planned for the extraction with intact non-metallic crown
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darya Dabiri, DMD, MS, Principal Investigator — University of Michigan
Locations (1):
- Oral and Maxiofacial Surgery Clinic, U of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oximetry Testing of Healthy Teeth and Those Requiring Removal: To assess the ability of pulse oximeter to assess the presence of pulse in teeth and to correlate pulse oximeter readings with conventional pulp testing measures including cold test, electrical pulp test, percussion and palpation testings, pulse oximeter will be used with a special holding frame, for 15-30 seconds.
  Note: the reading will not affect clinical practice; it is simply to gather data to see if pulse oximetry can facilitate diagnostic practices in the future
  Pulse Oximetry: Pulse Oximeter is being applied with a special holding tool to test the oximeter for its ability to measure pulpal blood flow, but no effect of the oximeter is being measured. Thus, to that degree the use is observational rather than interventional.
Period: Overall Study
Arm/Group | Oximetry Testing of Healthy Teeth and Those Requiring Removal
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oximetry Testing of Healthy Teeth and Those Requiring Removal
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 29
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Subjective Tooth Assessment: Number of Teeth With Normal and Abnormal Pulp
Description: Conventional subjective tooth assessments (percussion, palpation, cold, and electrical pulp testing) will be used for teeth that are planned for extraction and also upto 2-5 additional teeth in each participant. Pulp status is determined as "normal" or "abnormal" according to the classification system from the American Academy of Endodontics.
Time Frame: Single visit, less than one hour testing
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Groups:
- Oximetry Testing of Healthy Teeth and Those Requiring Removal: To assess the ability of pulse oximeter to assess the presence of pulse in teeth and to correlate pulse oximeter readings with conventional pulp testing measures including cold test, electrical pulp test, percussion and palpation testings, pulse oximeter will be used with a special holding frame, for 15-30 seconds.
  Note: the reading will not affect clinical practice; it is simply to gather data to see if pulse oximetry can facilitate diagnostic practices in the future. Pulse Oximetry: Pulse Oximeter is being applied with a special holding tool to test the oximeter for its ability to measure pulpal blood flow, but no effect of the oximeter is being measured.
Arm/Group | Oximetry Testing of Healthy Teeth and Those Requiring Removal
Number analyzed (Participants) | 29
Number analyzed (Teeth) | 143
Teeth
  Normal Pulp | 111
  Abnormal Pulp | 32

2. Secondary Outcome: Objective Tooth Assessment: Pulse Oximetry Reading for Selected Teeth
Description: Objective plural blood flow measurements will be used for teeth that are planned for extraction and also up to 2-5 additional teeth in each participant. Average objective plural blood flow was determined by pulse oximetry-reading for selected teeth (measured as SpO2).
Time Frame: Single visit, less than one hour testing
Measure: Mean (Standard Deviation); unit: Percentage of saturation
Units Other Than Participants: Teeth
Arm/Group | Oximetry Testing of Healthy Teeth and Those Requiring Removal
Number analyzed (Participants) | 29
Number analyzed (Teeth) | 143
Percentage of saturation | 87.9 (11.8)
Statistical Analysis 1: Comparison: Oximetry Testing of Healthy Teeth and Those Requiring Removal; Test type: Other; p = 0.92, ANOVA; Correlation Coefficient = 0.01

ADVERSE EVENTS:
Time Frame: Through study completion an average of one day
Arm/Group | Oximetry Testing of Healthy Teeth and Those Requiring Removal
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT03578549/Prot_SAP_001.pdf